CLINICAL TRIAL: NCT00478335
Title: Pharmacologic Treatment of Congenital Nephrogenic Diabetes Insipidus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-0588
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Nephrogenic Diabetes Insipidus
Keywords: congenital nephrogenic diabetes insipidus; polyuria; urine osmolality; aquaporin-2; vasopressin V2 receptor
MeSH Terms: conditions — Diabetes Insipidus, Nephrogenic; Polyuria | interventions — Sildenafil Citrate; Calcitonin; salmon calcitonin; amiloride, hydrochlorothiazide drug combination; Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Therapy (Experimental): 4-day treatment with hydrochlorothiazide/amiloride, indomethacin, calcitonin, sildenafil
  Interventions: Drug: sildenafil; Drug: calcitonin; Drug: hydrochlorothiazide/amiloride; Drug: indomethacin
- Placebo Control (Placebo Comparator): 4-day treatment with hydrochlorothiazide/amiloride, indomethacin, placebo for calcitonin, placebo for sildenafil
  Interventions: Drug: hydrochlorothiazide/amiloride; Drug: indomethacin; Drug: Placebo for sildenafil; Drug: placebo for calcitonin

INTERVENTIONS:
Drug: sildenafil — 25 mg quaque die (QD) or 50 mg QD x 4 days based on subject weight
  Other Names: Viagra
  Arms: Active Therapy
Drug: calcitonin — one nasal spray daily for 4 days
  Other Names: Miacalcic
  Arms: Active Therapy
Drug: hydrochlorothiazide/amiloride — 25 mg/2.5 mg BID or 50 mg/5 mg BID x 8 days depending on subject weight
  Other Names: Moduret, Moduretic
Drug: indomethacin — 50 mg QD or 50 mg BID x 8 days depending on subject weight
  Other Names: Indocin
Drug: Placebo for sildenafil — one tablet daily for 4 days
  Arms: Placebo Control
Drug: placebo for calcitonin — one nasal spray daily
  Arms: Placebo Control

SUMMARY:
The purpose of this research study is to determine if two investigational medications will be more effective in decreasing urine output than the currently available and routinely used medications in patients with congenital nephrogenic diabetes insipidus (NDI).

DETAILED DESCRIPTION:
The study involves the use of the investigational medications sildenafil and calcitonin. These medications have shown promise as treatment for NDI in laboratory (non-human) studies but have not been used for treatment of NDI in humans. At this time, there is no guarantee that these investigational medications will provide additional benefit to people with NDI.

The study is open to males, between the ages of 5 and 25 years who have been diagnosed with Nephrogenic diabetes insipidus (NDI) and who have normal kidney and bladder function. A total of 40 patients with NDI will be enrolled in the study. The study will involve two outpatient clinic visits, followed by a 9-night hospital stay, followed by a final follow-up outpatient clinic visit. All visits will take place within a 20-day time period.

At the first clinic visit, blood and urine testing for kidney and liver function and blood count will be performed. If the genetic alteration which causes your NDI has not been previously identified, blood for DNA testing will also be obtained. If a kidney and bladder ultrasound has not been performed in the past 6 months, it will be obtained. The ultrasound is to make sure that there is no problem with drainage of urine from the kidneys and bladder. Subjects will be asked to fill out food preference questionnaires to use for planning of meals for the hospital stay. Subjects will be given containers to collect two consecutive 24-hour urine samples at home. These urine collections will help determine how well the subjects routine medicines are working to control their NDI.

At the second clinic visit, subjects will bring in the two 24-hour urine samples. Blood will again be collected for further testing of kidney function. Subjects will be given containers to collect another 24-hour urine just prior to the hospital visit.

The third visit requires hospital admission and will be scheduled at the study site closest to the subjects home (The Children's Hospital, Denver, Colorado; University of Aarhus, Denmark). For the hospital visit, subjects will need to stop their usual NDI medications for 48 hours prior to the visit. Subjects will perform another 24-hour urine collection on the day prior to your hospital admission. This urine sample will be turned in to the laboratory when you are admitted to the hospital for the research study. The length of the hospital stay is 10 days/9 nights. During the stay, subjects can expect to have their weight, heart rate, and blood pressure checked three times a day. All urine will be collected. Blood testing will be performed every other day. Subjects will need to eat the meals provided at the hospital; all meals will be provided according to a low-salt diet restriction. Subjects may drink fluids as desired but they will need to avoid caffeine-containing beverages and alcohol.

On the first day of the hospital stay, testing will be performed to confirm the diagnosis of NDI. This test involves administration of the medicine dDAVP (Desmopressin) through an IV catheter (into a vein) with collection of urine every 30 minutes for 4 hours. subjects will be randomized (like the toss of a coin) to receive either the investigational medication treatment for 4 days followed by the routine medication treatment for 4 days or vice versa. When subjects receive the routine medication treatment, they will receive placebos (inactive substances like a sugar pill) in place of the investigational medicines. In this way, neither the subject nor the investigator will know whether the subjects are receiving the investigational or the routine medication treatment first. Medicines will be given twice a day during the hospital stay. On the last day of the hospital stay, subjects will be instructed to resume their normal diet and medications.

At a final outpatient clinic visit, blood testing and urinalysis will be performed.

Potential benefits of participation include a no-cost health examination, laboratory studies, and an evaluation of current management of NDI. There is no cost for participation in this research study. No pay will be given to participants in this research study.

This research study has been approved by the ethical review boards of the following institutions: Colorado Multiple Institutional Review Board (#06-0588), Emory University Institutional Review Board (#729-2005), and the University of Aarhus (#20050183). Individuals who decide to take part in this research study will need to sign a specific consent form at a participating institution as well as a release for use of personal health information (HIPAA form).

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of Congenital Nephrogenic Diabetes Insipidus (CNDI)
* Age 5 to 25 years
* Normal kidney function
* Post-void residual urine < 200 ml (determined by bladder ultrasound)

Exclusion Criteria:

* Impaired kidney function
* Known urinary retention or bladder dysfunction
* High blood pressure
* Other significant chronic medical disease (e.g., heart failure, liver disease, etc.)
* Allergy to study drugs

Ages: 5 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Cadnapaphornchai, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado at Denver and Health Sciences Center, Aurora, Colorado, United States
- University of Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bichet DG. Nephrogenic diabetes insipidus. Adv Chronic Kidney Dis. 2006 Apr;13(2):96-104. doi: 10.1053/j.ackd.2006.01.006. PMID 16580609
- [Background] Fujiwara TM, Bichet DG. Molecular biology of hereditary diabetes insipidus. J Am Soc Nephrol. 2005 Oct;16(10):2836-46. doi: 10.1681/ASN.2005040371. Epub 2005 Aug 10. PMID 16093448
- [Background] Schrier RW, Cadnapaphornchai MA. Renal aquaporin water channels: from molecules to human disease. Prog Biophys Mol Biol. 2003 Feb;81(2):117-31. doi: 10.1016/s0079-6107(02)00049-4. PMID 12565698
- [Background] Schrier RW, Cadnapaphornchai MA, Umenishi F. Water-losing and water-retaining states: role of water channels and vasopressin receptor antagonists. Heart Dis. 2001 May-Jun;3(3):210-4. doi: 10.1097/00132580-200105000-00014. PMID 11975794
- [Background] Nielsen S, Kwon TH, Frokiaer J, Agre P. Regulation and dysregulation of aquaporins in water balance disorders. J Intern Med. 2007 Jan;261(1):53-64. doi: 10.1111/j.1365-2796.2006.01760.x. PMID 17222168
- [Background] Kotnik P, Nielsen J, Kwon TH, Krzisnik C, Frokiaer J, Nielsen S. Altered expression of COX-1, COX-2, and mPGES in rats with nephrogenic and central diabetes insipidus. Am J Physiol Renal Physiol. 2005 May;288(5):F1053-68. doi: 10.1152/ajprenal.00114.2004. Epub 2005 Jan 11. PMID 15644490
- [Background] Nielsen S, Frokiaer J, Marples D, Kwon TH, Agre P, Knepper MA. Aquaporins in the kidney: from molecules to medicine. Physiol Rev. 2002 Jan;82(1):205-44. doi: 10.1152/physrev.00024.2001. PMID 11773613
- [Background] Bouley R, Pastor-Soler N, Cohen O, McLaughlin M, Breton S, Brown D. Stimulation of AQP2 membrane insertion in renal epithelial cells in vitro and in vivo by the cGMP phosphodiesterase inhibitor sildenafil citrate (Viagra). Am J Physiol Renal Physiol. 2005 Jun;288(6):F1103-12. doi: 10.1152/ajprenal.00337.2004. Epub 2005 Jan 11. PMID 15644488
- See also: Nephrogenic Diabetes Insipidus Foundation — http://www.ndif.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental First Then Standard: Experimental phase: 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), calcitonin (one nasal spray daily for 4 days), sildenafil (25 mg quaque die (QD) or 50 mg QD x 4 days based on subject weight).
  Followed by 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), Placebo for calcitonin (one nasal spray daily), Placebo for sildenafil (1 tablet daily).
- Standard First Then Experimental: 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), Placebo for calcitonin (one nasal spray daily), Placebo for sildenafil (1 tablet daily).
  Followed by 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), calcitonin (one nasal spray daily for 4 days), sildenafil (25 mg quaque die (QD) or 50 mg QD x 4 days based on subject weight).
Period: Period 1 (4 Days)
Arm/Group | Experimental First Then Standard | Standard First Then Experimental
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Period 2 (4 Days)
Arm/Group | Experimental First Then Standard | Standard First Then Experimental
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: crossover
Groups:
- Experimental First Then Standard: 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), calcitonin (one nasal spray daily for 4 days), sildenafil (25 mg quaque die (QD) or 50 mg QD x 4 days based on subject weight).
  Followed by 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), Placebo for calcitonin (one nasal spray daily), Placebo for sildenafil (1 tablet daily).
- Total: Total of all reporting groups
Arm/Group | Experimental First Then Standard | Standard First Then Experimental | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 24h Urine Volume
Description: urine volume in mL/d
Time Frame: 4-days
Measure: Mean (Standard Deviation); unit: urine volume in mL/d
Groups:
- Experimental First Then Standard: 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), calcitonin (one nasal spray daily for 4 days), sildenafil (25 mg quaque die (QD) or 50 mg QD x 4 days based on subject weight).
  Followed by 4-day treatment with hydrochlorothiazide/amiloride (25 mg/2.5 mg BID or 50 mg/5 mg BID based on subject weight), indomethacin (50 mg QD or 50 mg BID based on subject weight), Placebo for calcitonin (one nasal spray daily), Placebo for sildenafil (1 tablet daily).
  on subject weight
Arm/Group | Experimental First Then Standard | Standard First Then Experimental
Number analyzed (Participants) | 2 | 2
urine volume in mL/d
  Period 1 | 6475 (742) | 4178 (590)
  Period 2 | 6652 (1305) | 4188 (1679)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Description: Adverse events were evaluated based on clinical course and via use of systematic written survey to all participants
Arm/Group | Experimental First Then Standard | Standard First Then Experimental
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes